CLINICAL TRIAL: NCT01408121
Title: African-American Pharmacogenetics
Acronym: AA Genetic
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: AA Genetic
Record Dates: First submitted 2011-07-29; First posted 2011-08-03 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Acute Coronary Syndrome
Keywords: Platelet reactivity; Genotyping
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Genotype

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- African-American on clopidogrel
  Interventions: Other: Genotyping and platelet reactivity testing with the VerifyNow P2Y12 assay
- African-American on prasugrel
  Interventions: Other: Genotyping and platelet reactivity testing with the VerifyNow P2Y12 assay
- Caucasian on clopidogrel
  Interventions: Other: Genotyping and platelet reactivity testing with the VerifyNow P2Y12 assay
- Caucasian on prasugrel
  Interventions: Other: Genotyping and platelet reactivity testing with the VerifyNow P2Y12 assay

INTERVENTIONS:
Other: Genotyping and platelet reactivity testing with the VerifyNow P2Y12 assay — All patients will undergo genotyping and platelet reactivity testing with the VerifyNow P2Y12 assay, at least 6 hours after receiving a thienopyridine loading dose but before hospital discharge.

SUMMARY:
This is a genetic and platelet reactivity study of African-American versus Caucasian patients undergoing percutaneous coronary intervention and receiving clopidogrel or prasugrel. The investigators aim is twofold: to describe differences in allele frequencies between African-Americans and Caucasians, and to explore associations of platelet reactivity and genetic polymorphisms in these two groups.

DETAILED DESCRIPTION:
The investigators propose a pharmacogenetic cohort study of 100 African-American versus 100 Caucasian patients presenting with an acute coronary syndrome, receiving clopidogrel or prasugrel and undergoing PCI. The study will have four arms: African-American on clopidogrel; African-American on prasugrel; Caucasian on clopidogrel; and Caucasian on prasugrel. All patients will undergo genotyping and platelet reactivity testing with the VerifyNow P2Y12 assay, at least 6 hours after receiving a thienopyridine loading dose, but before hospital discharge. All patients will be treated with aspirin 325 mg/day as well.

Race determination will be based on a patient's self-report, but patients enrolled in the trial must also report that all four of their grandparents were of the same race as theirs. Other races (Asian, Native American, et al) will be excluded from this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18 or older, of both genders
2. Presenting with an ACS, defined as at least two of the following:

   * symptoms consistent with myocardial ischemia;
   * ST segment elevation or depression of at least 1 mm in 2 or more contiguous leads on EKG;
   * a cardiac troponin I level above upper limit of normal.
3. Self-reported African-american or Caucasian race

   a. all 4 grandparents of same race
4. No contraindications to prasugrel therapy.
5. Patient is scheduled for, or has already undergone, PCI.

Exclusion Criteria:

1. Known allergies to aspirin, clopidogrel, or prasugrel.
2. Patient known to be pregnant or lactating.
3. Patient with known history of bleeding diathesis or currently active bleeding.
4. Platelet count <100,000/mm at the time of enrollment.
5. Hematocrit <25% at the time of enrollment.
6. On warfarin therapy at the time of PCI, or patient likely to require warfarin therapy post-PCI.
7. Received fibrinolytics within the past 48 hours.
8. Received a glycoprotein IIb/IIIa inhibitor within the past 48 hours, or if such a strategy for PCI involving a glycoprotein IIb/IIIa inhibitor is planned.
9. Taking maintenance thienopyridine therapy in the previous 5 days.
10. Known blood transfusion within the preceding 10 days.
11. Patients treated with non-steroidal anti-inflammatory drugs (NSAIDS) within the previous 5 days.
12. Patients with known chronic liver disease.
13. Age greater than 75 years
14. Body weight less than 60 kg
15. History of stroke or transient ischemic attack
16. Surgery planned within 1 month
17. Patient likely to require coronary artery bypass grafting
18. Any significant medical condition that, in the investigator's opinion, may interfere with the patient's optimal participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: African-american versus Caucasian patients undergoing percutaneous coronary intervention and receiving clopidogrel or prasugrel.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-11; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Distribution of CYP polymorphisms | During hospital stay; average hospital stay is less than 48 hours
  CYP polymorphisms will be classified by their known effects upon enzyme function, using the consensus star-allele nomenclature. More specifically, patients will be classified as a "poor metabolizer" if they possess at least one CYP allele known to be associated with reduced function of that particular CYP enzyme. Allele frequencies will then be compared between African-american and Caucasian patients.

SECONDARY OUTCOMES:
Platelet reactivity | During hospital stay; average hospital stay is less than 48 hours
  The secondary exploratory objective is to assess for associations between "poor metabolizer" CYP genotypes and the levels of post-thienopyridine platelet reactivity.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States